CLINICAL TRIAL: NCT04730869
Title: Feasibility, Safety, and Efficacy of a Metabolic Therapy Program in Conjunction With Standard Treatment for Glioblastoma
Brief Title: Metabolic Therapy Program In Conjunction With Standard Treatment For Glioblastoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Waikato Hospital (Other)
Collaborators: Wellington Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD020132; U1111-1262-0203 (Other: International Clinical Trials Registry Platform); Grant #321 (Other Grant/Funding Number: Waikato Medical Research Foundation)
Record Dates: First submitted 2020-12-22; First posted 2021-01-29 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Glioblastoma
Keywords: cancer; glioblastoma; metabolic therapy; fasting; ketogenic diet
MeSH Terms: conditions — Glioblastoma; Neoplasms; Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standard treatment in conjunction with MTP (Experimental): Standard:
  * Concurrent chemoradiation - Radiation (60-Gy in 30 fractions over 6 weeks) with daily oral temozolomide.
  * Adjuvant chemotherapy - Daily oral temozolomide (5 days per 4-week cycle, starting 4 weeks after completion of chemoradiation, with at least 6 cycles intended).
  MTP:
  - Two 5-day fasts (allowing water, salt, tea, coffee, and a magnesium supplement) during chemoradiation followed by a 5-day fast during each adjuvant chemotherapy cycle, with a time-restricted modified ketogenic diet (one or two 1-hour eating windows per day, allowing oils, meats, vegetables, nuts, seeds, limited berries, and a multivitamin) between fasts.
  Interventions: Other: Standard Treatment Plus Metabolic Therapy Program

INTERVENTIONS:
Other: Standard Treatment Plus Metabolic Therapy Program — See description under "Arms."

SUMMARY:
Glioblastoma (GBM), a very aggressive brain tumour, is one of the most malignant of all cancers and is associated with a poor prognosis. The majority of GBM cells display damaged mitochondria (the "batteries" of cells), so they rely on an alternate method for producing energy called the Warburg Effect, which relies nearly exclusively on glucose (in contrast, normal cells can use other molecules, such as fatty acids and fat-derived ketones, for energy). Metabolic interventions, such as fasting and ketogenic diets, target cancer cell metabolism by enhancing mitochondria function, decreasing blood glucose levels, and increasing blood ketone levels, creating an advantage for normal cells but a disadvantage for cancer cells. Preliminary experience at Waikato Hospital has shown that a metabolic therapy program (MTP) utilizing fasting and ketogenic diets is feasible and safe in people with advanced cancer, and may provide a therapeutic benefit. We aim to determine whether using an MTP concurrently with standard oncological treatment (chemoradiation followed by adjuvant chemotherapy) is feasible and safe in patients with GBM, and has treatment outcomes consistent with greater overall treatment efficacy than in published trials.

DETAILED DESCRIPTION:
Gliomas are tumours that originate from glial cells in the central nervous system. The most common histological subtype is GBM, which accounts for nearly 50% of all malignant brain tumours. Despite aggressive multimodal treatment, the median survival for GBM is poor (8-15 months).

Although cancer is regarded as a genetic disease, it may be perceived as a metabolic disorder. The majority of human cancers, including GBM, display low numbers of mitochondria, most of which are structurally damaged, resulting in defective cell respiration. To compensate, cancer cells greatly increase their uptake of glucose, which is fermented (regardless of oxygen concentration, a process known as the Warburg Effect) to generate energy. Cancer cells also rely on increased growth signaling pathways involving insulin, insulin-like growth factor-1, and mammalian target of rapamycin to support their unbridled growth and proliferation. Cancer cells may therefore be vulnerable to interventions that selectively target their abnormal metabolism.

Metabolic interventions, such as fasting and ketogenic diets, target cancer cell metabolism and may be effective alongside standard treatments in advanced cancers. Fasting is a voluntary abstinence from food and drink for a controlled period of time (typically, 12 hours to 3 weeks in humans), whereas ketogenic diets are high-fat, adequate-protein, low-carbohydrate diets that stimulate the body to create a fasting-like metabolic state. Fasting and ketogenic diets stimulate mitochondria biogenesis, decrease blood glucose, increase liver production of fat-derived ketones (which serve as a major alternative energy source for most normal cells within the body, but cannot be utilized by cancer cells), and decrease growth factor availability. Thus, fasting and ketogenic diets provide an advantage for normal cells but a disadvantage to cancer cells by enhancing mitochondria biogenesis and function, depriving cancer cells of their major fuel, and creating a cell environment unfavourable for unbridled growth and proliferation.

Preliminary experience at Waikato Hospital has shown that a metabolic therapy program (MTP) consisting of fasting and/or a ketogenic diet is feasible, safe, and may be effective in patients with advanced cancer, including GBM. In a recent case report, a metabolic strategy (7-day fast every 1-2 months, with a ketogenic diet between fasts) resulted in the near-complete regression of a stage IVA metastatic thymoma after 2 years. Moreover, we are currently observing 8 glioblastoma patients who voluntarily consented to undergo fasting and ketogenic diet therapy in a manner similar to what we propose to use in this study; at an average of 4-5 months, all patients have completed the fasts and adhered to their ketogenic diet, experiencing only mild adverse effects.

On this background, we aim to determine whether using an MTP concurrently with standard oncological treatment (chemoradiation followed by adjuvant chemotherapy) is feasible and safe, and has treatment outcomes consistent with greater overall treatment efficacy than in published trials, in patients with GBM.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or greater.
2. Newly-diagnosed histologically-confirmed GBM.
3. ECOG Performance Status 0-2.
4. Planned for 6 weeks of standard chemoradiation for GBM.
5. If receiving dexamethasone, the dose must be ≤ 4 mg daily (and not increasing) upon commencement of the MTP.

Exclusion Criteria:

1. Ineligible for standard treatment for GBM due to poor performance status, co-morbidities, or inability to give informed consent.
2. Type 1 diabetes.
3. A medical or psychiatric disorder that, in the opinion of the investigators, would make it unlikely that the patient could adhere to the MTP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
Mean daily blood glucose-to-ketone ratio during chemoradiation | 9 weeks
  Proportion of patients able to sustain functional ketosis (defined as a mean daily blood glucose-to-ketone ratio of ≤6) during chemoradiation (defined as the beginning of the first fast through to 3 weeks following completion of chemoradiation)

SECONDARY OUTCOMES:
Mean daily blood glucose-to-ketone ratio during adjuvant chemotherapy | 24 weeks
  Proportion of patients able to sustain functional ketosis during adjuvant chemotherapy (defined as the beginning of the first adjuvant chemotherapy fast through to completion of adjuvant chemotherapy)
Mean daily blood glucose-to-ketone ratio during the MTP, calculated separately on fasting and ketogenic diet days | 33 weeks
  Proportion of patients able to sustain functional ketosis during the MTP (defined as the beginning of chemoradiation through to the end of adjuvant chemotherapy), calculated separately each fasting and ketogenic diet phase
Change in weight | 33 weeks
  Weight (kg)
Safety as measured by National Cancer Institute Common Terminology Criteria for Adverse Events (version 4) | After each week (7 days) during chemoradiation, then after cycle 1 (28 days) of adjuvant chemotherapy, then after every 2 cycles (56 days) of adjuvant chemotherapy
  Number of adverse events (of any grade)
Change in performance status as measured by Eastern Cooperative Oncology Group Performance Status scale | After each week (7 days) during chemoradiation, then after cycle 1 (28 days) of adjuvant chemotherapy, then after every 2 cycles (56 days) of adjuvant chemotherapy
  Eastern Cooperative Oncology Group Performance Status scale (scores range from 0 to 5, with higher scores indicating lower performance status)
Change in leisure/exercise activity as measured by Godin Leisure-Time Exercise questionnaire | After each week (7 days) during chemoradiation, then after cycle 1 (28 days) of adjuvant chemotherapy, then after every 2 cycles (56 days) of adjuvant chemotherapy
  Godin Leisure-Time Exercise questionnaire (scores range from 0 to no maximum, with higher scores indicating higher leisure/exercise activity)
Change in quality of life as measured by Functional Assessment of Cancer Therapy - Brain questionnaire | After each week (7 days) during chemoradiation, then after cycle 1 (28 days) of adjuvant chemotherapy, then after every 2 cycles (56 days) of adjuvant chemotherapy
  Functional Assessment of Cancer Therapy - Brain questionnaire (scores range from 0 to 200, with higher scores indicating higher quality of life)
Progression-free survival | From date of biopsy-confirmed diagnosis to date of first documented progression, whichever came first, up to 33 weeks
  Progression-free survival
Overall survival | From date of biopsy-confirmed diagnosis to date of death from any cause, whichever came first, up to 33 weeks
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Matthew CL Phillips, FRACP, Principal Investigator — Waikato Hospital
Locations (1):
- Waikato Hospital, Hamilton, Waikato Region, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request for research purposes only, de-identified patient data may be shared with other investigators.
Supporting Information: Study Protocol
Time Frame: Starting immediately upon publication.
Access Criteria: Upon reasonable request for research purposes.